CLINICAL TRIAL: NCT00153855
Title: Structural Brain Abnormalities in Children Born Prematurely: New Detection Methods and Clinical-Pathological Correlates
Status: Terminated | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Boston Children's Hospital (Other); Children's Mercy Hospital Kansas City (Other)
Other Study IDs: 2004-6-3818
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Infant, Premature; Brain Injuries
Keywords: etiology; pathology
MeSH Terms: conditions — Premature Birth; Brain Injuries

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of the study is to detect structural brain changes using MRI and to correlate these findings with neurodevelopmental assessments in two-year old children previously enrolled in the NIH sponsored trial of inhaled Nitric Oxide (iNO) for the prevention of Chronic Lung Disease in preterm ventilated infants. It is hypothesized that this imaging will identify children with previously undiagnosed brain abnormalities and that the presence of structural abnormalities will be associated with deficits in motor, cognitive, and neurosensory development.

DETAILED DESCRIPTION:
Infants born prematurely are at significant risk for hemorrhagic and ischemic brain injury. Despite improved survival rates among this population in recent years, these forms of brain injury remain frequent and have considerable consequences. Periventricular leukomalacia (PVL), a disease characterized by necrosis of the cerebral white matter in a characteristic distribution, is one of the most common types of brain injury seen in premature infants. MRI technology now allows for better anatomical resolution resulting in improvements in diagnostic accuracy. The current standard practice is not to perform routine MRI examinations on premature infants, nor is it routine to perform surveillance brain imaging in children after leaving the NICU. In their 2002 Practice Parameter for neuroimaging in the neonate, the American Academy of Neurology and the Practice Committee of the Child Neurology Society acknowledge the superiority of MRI in detection of brain lesions in premature infants, but fall short of recommending routine MRI scanning on the basis of a lack of information correlating MRI findings to neurodevelopmental outcomes. We now have a unique opportunity to help provide such information.

ELIGIBILITY:
Inclusion Criteria:

* must be participants in trial (NHLBI-UO1-HL62514-05A1 and FDA IND # 58,146 - Roberta A Ballard PI) of inhaled Nitric Oxide (iNO) for the prevention of Chronic Lung Disease in preterm ventilated infants
* gestational age between 24 months and 27 months

Exclusion Criteria:

* history of allergy to sedation agents
* medical conditions which may pose a threat to airway integrity (i.e., Pierre-Robin sequence, intercurrent respiratory illness)
* other conditions which may otherwise place subjects at increased risk for complications from sedation and MRI examination

Ages: 24 Months to 27 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50
Dates: Start 2005-01; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Roberta A Ballard, M.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Stevenson DK, Wright LL, Lemons JA, Oh W, Korones SB, Papile LA, Bauer CR, Stoll BJ, Tyson JE, Shankaran S, Fanaroff AA, Donovan EF, Ehrenkranz RA, Verter J. Very low birth weight outcomes of the National Institute of Child Health and Human Development Neonatal Research Network, January 1993 through December 1994. Am J Obstet Gynecol. 1998 Dec;179(6 Pt 1):1632-9. doi: 10.1016/s0002-9378(98)70037-7. PMID 9855609
- [Background] Volpe JJ. Brain injury in the premature infant: overview of clinical aspects, neuropathology, and pathogenesis. Semin Pediatr Neurol. 1998 Sep;5(3):135-51. doi: 10.1016/s1071-9091(98)80030-2. PMID 9777673
- [Background] Hack M, Fanaroff AA. Outcomes of children of extremely low birthweight and gestational age in the 1990s. Semin Neonatol. 2000 May;5(2):89-106. doi: 10.1053/siny.1999.0001. PMID 10859704
- [Background] Bhutta AT, Cleves MA, Casey PH, Cradock MM, Anand KJ. Cognitive and behavioral outcomes of school-aged children who were born preterm: a meta-analysis. JAMA. 2002 Aug 14;288(6):728-37. doi: 10.1001/jama.288.6.728. PMID 12169077
- [Background] Sie LT, van der Knaap MS, van Wezel-Meijler G, Taets van Amerongen AH, Lafeber HN, Valk J. Early MR features of hypoxic-ischemic brain injury in neonates with periventricular densities on sonograms. AJNR Am J Neuroradiol. 2000 May;21(5):852-61. PMID 10815660
- [Background] Inder TE, Huppi PS, Warfield S, Kikinis R, Zientara GP, Barnes PD, Jolesz F, Volpe JJ. Periventricular white matter injury in the premature infant is followed by reduced cerebral cortical gray matter volume at term. Ann Neurol. 1999 Nov;46(5):755-60. doi: 10.1002/1531-8249(199911)46:53.0.co;2-0. PMID 10553993
- [Background] Olsen P, Paakko E, Vainionpaa L, Pyhtinen J, Jarvelin MR. Magnetic resonance imaging of periventricular leukomalacia and its clinical correlation in children. Ann Neurol. 1997 Jun;41(6):754-61. doi: 10.1002/ana.410410611. PMID 9189036
- [Background] Inder TE, Wells SJ, Mogridge NB, Spencer C, Volpe JJ. Defining the nature of the cerebral abnormalities in the premature infant: a qualitative magnetic resonance imaging study. J Pediatr. 2003 Aug;143(2):171-9. doi: 10.1067/S0022-3476(03)00357-3. PMID 12970628
- [Background] Huppi PS, Murphy B, Maier SE, Zientara GP, Inder TE, Barnes PD, Kikinis R, Jolesz FA, Volpe JJ. Microstructural brain development after perinatal cerebral white matter injury assessed by diffusion tensor magnetic resonance imaging. Pediatrics. 2001 Mar;107(3):455-60. doi: 10.1542/peds.107.3.455. PMID 11230582
- [Background] Huppi PS, Maier SE, Peled S, Zientara GP, Barnes PD, Jolesz FA, Volpe JJ. Microstructural development of human newborn cerebral white matter assessed in vivo by diffusion tensor magnetic resonance imaging. Pediatr Res. 1998 Oct;44(4):584-90. doi: 10.1203/00006450-199810000-00019. PMID 9773850
- [Background] Hoon AH Jr, Lawrie WT Jr, Melhem ER, Reinhardt EM, Van Zijl PC, Solaiyappan M, Jiang H, Johnston MV, Mori S. Diffusion tensor imaging of periventricular leukomalacia shows affected sensory cortex white matter pathways. Neurology. 2002 Sep 10;59(5):752-6. doi: 10.1212/wnl.59.5.752. PMID 12221171
- [Background] Miller SP, Vigneron DB, Henry RG, Bohland MA, Ceppi-Cozzio C, Hoffman C, Newton N, Partridge JC, Ferriero DM, Barkovich AJ. Serial quantitative diffusion tensor MRI of the premature brain: development in newborns with and without injury. J Magn Reson Imaging. 2002 Dec;16(6):621-32. doi: 10.1002/jmri.10205. PMID 12451575
- [Background] Inder TE, Volpe JJ. Mechanisms of perinatal brain injury. Semin Neonatol. 2000 Feb;5(1):3-16. doi: 10.1053/siny.1999.0112. PMID 10802746
- [Background] Melhem ER, Hoon AH Jr, Ferrucci JT Jr, Quinn CB, Reinhardt EM, Demetrides SW, Freeman BM, Johnston MV. Periventricular leukomalacia: relationship between lateral ventricular volume on brain MR images and severity of cognitive and motor impairment. Radiology. 2000 Jan;214(1):199-204. doi: 10.1148/radiology.214.1.r00dc35199. PMID 10644124
- [Background] Ment LR, Bada HS, Barnes P, Grant PE, Hirtz D, Papile LA, Pinto-Martin J, Rivkin M, Slovis TL. Practice parameter: neuroimaging of the neonate: report of the Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. Neurology. 2002 Jun 25;58(12):1726-38. doi: 10.1212/wnl.58.12.1726. PMID 12084869
- [Background] Early compared with delayed inhaled nitric oxide in moderately hypoxaemic neonates with respiratory failure: a randomised controlled trial. The Franco-Belgium Collaborative NO Trial Group. Lancet. 1999 Sep 25;354(9184):1066-71. PMID 10509497
- [Background] Bennett AJ, Shaw NJ, Gregg JE, Subhedar NV. Neurodevelopmental outcome in high-risk preterm infants treated with inhaled nitric oxide. Acta Paediatr. 2001 May;90(5):573-6. PMID 11430720
- [Background] Cheung PY, Peliowski A, Robertson CM. The outcome of very low birth weight neonates (</=1500 g) rescued by inhaled nitric oxide: neurodevelopment in early childhood. J Pediatr. 1998 Dec;133(6):735-9. doi: 10.1016/s0022-3476(98)70142-8. PMID 9842035
- [Background] Kinsella JP, Walsh WF, Bose CL, Gerstmann DR, Labella JJ, Sardesai S, Walsh-Sukys MC, McCaffrey MJ, Cornfield DN, Bhutani VK, Cutter GR, Baier M, Abman SH. Inhaled nitric oxide in premature neonates with severe hypoxaemic respiratory failure: a randomised controlled trial. Lancet. 1999 Sep 25;354(9184):1061-5. doi: 10.1016/s0140-6736(99)03558-8. PMID 10509496
- [Background] Rosenberg AA, Kennaugh JM, Moreland SG, Fashaw LM, Hale KA, Torielli FM, Abman SH, Kinsella JP. Longitudinal follow-up of a cohort of newborn infants treated with inhaled nitric oxide for persistent pulmonary hypertension. J Pediatr. 1997 Jul;131(1 Pt 1):70-5. doi: 10.1016/s0022-3476(97)70126-4. PMID 9255194
- [Background] Subhedar NV, Ryan SW, Shaw NJ. Open randomised controlled trial of inhaled nitric oxide and early dexamethasone in high risk preterm infants. Arch Dis Child Fetal Neonatal Ed. 1997 Nov;77(3):F185-90. doi: 10.1136/fn.77.3.f185. PMID 9462187
- [Background] Schreiber MD, Gin-Mestan K, Marks JD, Huo D, Lee G, Srisuparp P. Inhaled nitric oxide in premature infants with the respiratory distress syndrome. N Engl J Med. 2003 Nov 27;349(22):2099-107. doi: 10.1056/NEJMoa031154. PMID 14645637